CLINICAL TRIAL: NCT01303952
Title: Therapy for Chronic Cold Agglutinin Disease: A Prospective, Non-Randomized Multi-Center Study Demonstrating the Efficacy of Terminal Complement Inhibition in Patients With Cold Agglutinin Disease Using Eculizumab
Brief Title: Therapy of Chronic Cold Agglutinin Disease With Eculizumab
Acronym: DECADE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Alexander Roeth, MD, MD, University Hospital, Essen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAD01; 2009-016966-97 (EudraCT Number)
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Cold Agglutinin Disease
Keywords: cold agglutinin disease; hemolysis; eculizumab; terminal complement inhibition
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Hemolysis | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eculizumab (Experimental)
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Weekly treatment with eculizumab (600 mg) via IV infusion for 4 doses followed the next week by eculizumab (900 mg) IV infusion and maintenance treatment with Eculizumab (900 mg) via IV infusion every other week for 21 weeks

SUMMARY:
Evaluation of the efficacy and safety of eculizumab in symptomatic or transfusion-dependent patients with untreated or refractory hemolytic cold agglutinin disease(CAD)

ELIGIBILITY:
Inclusion Criteria:

* Individuals at least 18 years of age
* Diagnosis of CAD defined by the combination of chronic hemolysis, cold agglutinin titer (IgM or IgA) >64 at 4°C, positive direct antiglobulin test (DAT) when performed with polyspecific antiserum, negative (or only weakly positive) anti-IgG, and strongly positive with anti-C3d
* LDH level > 2 x upper limit of normal (ULN)
* Clinical symptoms requiring treatment, such as anemia, anemia-related symptoms or hemolysis-related symptoms
* Sufficient supplementation of iron, folic acid and vitamin B12 prior to treatment phase
* Patient must be willing and able to give written informed consent;
* Patients must be vaccinated against N. meningitidis at least 14 days prior treatment
* Patient must avoid conception during the trial using a method that is most appropriate for their physical state and culture

Exclusion Criteria:

* Active aggressive lymphoma requiring therapy or an active non-lymphatic malignant disease other than basal cell carcinoma or CIS of the cervix
* Liver disease with elevated LDH
* Absolute neutrophil count < 500/µL
* Presence or suspicion of active bacterial or viral infection, in the opinion of the Investigator, at treatment start or severe recurrent bacterial infections
* Participation in any other investigational drug trial or exposure to other investigational agent, device, or procedure within 30 days prior to screening period
* Pregnant, breast-feeding, or intending to conceive during the course of the study, including the Post-treatment Phase
* History of bone marrow/stem cell transplantation
* Inability to cooperate or any condition that, in the opinion of the investigator, could increase the patient's risk by participating in the study or confound the outcome of the study
* Hypersensitivity to eculizumab, to murine proteins or to one of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
LDH | From baseline to 26 weeks
  Primary endpoint for this study is: lactate dehydrogenase (LDH) in U/l change from baseline to 26 weeks

SECONDARY OUTCOMES:
Transfusion avoidance | From baseline to 26 weeks
PRBC units transfused | From baseline to 26 weeks
Change in hemoglobin levels | From baseline to 26 weeks
Haptoglobin | From baseline to 26 weeks
Hemopexin | From baseline to 26 weeks
Free hemoglobin | From baseline to 26 weeks
Reticulocytes | From baseline to 26 weeks
SF-36v2 QLQ | From baseline to 26 weeks
FACIT-F SCALE version 4 | From baseline to 26 weeks
Six-Minute Walk Test | From baseline to 26 weeks
Circulatory symptoms | From baseline to 26 weeks
Thrombosis record | From baseline to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Roeth, MD, Principal Investigator — Department of Hematology, University Hospital Essen
Locations (1):
- Department of Hematology, University Hospital Essen, Essen, Germany

REFERENCES:
- [Background] Roth A, Huttmann A, Rother RP, Duhrsen U, Philipp T. Long-term efficacy of the complement inhibitor eculizumab in cold agglutinin disease. Blood. 2009 Apr 16;113(16):3885-6. doi: 10.1182/blood-2009-01-196329. No abstract available. PMID 19372265
- [Background] Roth A, Duhrsen U. Cold agglutinin disease. Eur J Haematol. 2010 Jan 1;84(1):91. doi: 10.1111/j.1600-0609.2009.01320.x. Epub 2009 Jul 14. No abstract available. PMID 19614954
- [Derived] Roth A, Bommer M, Huttmann A, Herich-Terhurne D, Kuklik N, Rekowski J, Lenz V, Schrezenmeier H, Duhrsen U. Eculizumab in cold agglutinin disease (DECADE): an open-label, prospective, bicentric, nonrandomized phase 2 trial. Blood Adv. 2018 Oct 9;2(19):2543-2549. doi: 10.1182/bloodadvances.2018024190. PMID 30291112